CLINICAL TRIAL: NCT01142778
Title: An Open-Label, Randomized, Multicenter, Phase II, Non Comparative, Exploratory Study on Neoadjuvant Treatment With Trastuzumab Plus Docetaxel Plus Bevacizumab According to Positon Emission Tomography (PET) Value Modification in Patients With Early Stage HER2 Positive Breast Cancer
Brief Title: A Study of Bevacizumab Added to Trastuzumab Plus Docetaxel in the Neoadjuvant Setting in Participants With Early Stage HER2-Positive Breast Cancer
Acronym: AVATAXHER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML22229; 2009-013410-26 (EudraCT Number)
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Docetaxel; Trastuzumab; Surgical Procedures, Operative; Radiotherapy

ARMS (3):
- Trastuzumab, Docetaxel, and Bevacizumab (Experimental): Participants will receive 2 cycles of trastuzumab and docetaxel once every 3 weeks. Then, participants with a response of <70% will receive trastuzumab and docetaxel along with bevacizumab in Cycles 3 to 6. All participants will receive trastuzumab alone in Cycle 7, and will undergo surgery after Cycle 7 and between 4 and 6 weeks after the bevacizumab infusion in Cycle 6. After surgery, all participants will receive a further 11 cycles of trastuzumab plus radiotherapy with or without hormonal therapy as per site's standard practice, and will be followed for up to 5 years from start of neoadjuvant treatment.
  Interventions: Drug: Bevacizumab; Drug: Docetaxel; Drug: Trastuzumab; Procedure: Surgery; Radiation: Radiotherapy; Drug: Hormonal Therapy
- Trastuzumab and Docetaxel (Active Comparator): Participants will receive 2 cycles of trastuzumab and docetaxel once every 3 weeks. Then, participants with a response of <70% will receive trastuzumab and docetaxel in Cycles 3 to 6. All participants will receive trastuzumab alone in Cycle 7, and will undergo surgery after Cycle 7 and between 4 and 6 weeks after the study treatment perfusion in Cycle 6. After surgery, all participants will receive a further 11 cycles of trastuzumab plus radiotherapy with or without hormonal therapy as per site's standard practice, and will be followed for up to 5 years from start of neoadjuvant treatment.
  Interventions: Drug: Docetaxel; Drug: Trastuzumab; Procedure: Surgery; Radiation: Radiotherapy; Drug: Hormonal Therapy
- Trastuzumab and Docetaxel (Standard Regimen) (Active Comparator): Participants will receive 2 cycles of trastuzumab and docetaxel once every 3 weeks. Then, participants with a response of >/=70% will receive trastuzumab and docetaxel in Cycles 3 to 6. All participants will receive trastuzumab alone in Cycle 7, and will undergo surgery after Cycle 7 and between 4 and 6 weeks after the study treatment perfusion in Cycle 6. After surgery, all participants will receive a further 11 cycles of trastuzumab plus radiotherapy with or without hormonal therapy as per site's standard practice, and will be followed for up to 5 years from start of neoadjuvant treatment.
  Interventions: Drug: Docetaxel; Drug: Trastuzumab; Procedure: Surgery; Radiation: Radiotherapy; Drug: Hormonal Therapy

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab at a dose of 15 mg/kg will be administered as IV infusion over 90 minutes from Cycles 3-6 (1 Cycle=21 days).
  Other Names: Avastin
  Arms: Trastuzumab, Docetaxel, and Bevacizumab
Drug: Docetaxel — Docetaxel at a dose of 100 mg/m^2 will be administered as IV infusion from Cycles 1-6 (1 Cycle=21 days).
  Other Names: Taxotere
Drug: Trastuzumab — Trastuzumab will be administered as a loading dose of 8 mg/kg as IV infusion in Cycle 1, followed by subsequent dose of 6 mg/kg as IV infusion in Cycles 2 to 7, and during additional 11 cycles post surgery (1 Cycle=21 days).
  Other Names: Herceptin
Procedure: Surgery — All participants will undergo surgery (as per investigator's discretion) after Cycle 7 and between 4 and 6 weeks after the study treatment infusion in Cycle 6 (1 Cycle=21 days).
Radiation: Radiotherapy — All participants will receive radiotherapy starting about 4 to 8 weeks after surgery, and will last around 4 to 6 weeks as per site's standard practice.
Drug: Hormonal Therapy — Participants who are hormone receptors positive, will receive hormonal therapy after completion of radio therapy period as per investigator's discretion and site's standard practice.

SUMMARY:
This randomized study will assess the effect of adding bevacizumab to trastuzumab plus docetaxel in neoadjuvant therapy in participants with early stage human epidermal growth factor receptor 2 (HER2)-positive breast cancer. After 2 cycles of trastuzumab and docetaxel once every 3 weeks, participants with a response (change in standard uptake value [SUV]) of less than (<) 70 percent (%) on Positron Emission Tomography (PET) will be randomized in a 2:1 ratio to receive Cycles 3 to 6 of trastuzumab (6 milligrams per kilogram [mg/kg]) and docetaxel (100 milligrams per square meter [mg/m^2]) with or without bevacizumab (15 mg/kg). Participants with a response of greater than or equal to (>/=) 70% will receive trastuzumab plus docetaxel in Cycles 3 to 6. All participants will receive trastuzumab alone in Cycle 7, and will undergo surgery (as per investigator's discretion) after Cycle 7 and between 4 and 6 weeks after the treatment perfusion of Cycle 6. After surgery, all participants will receive a further 11 cycles of trastuzumab plus radiotherapy (starting from 4-8 weeks after surgery during 4-6 weeks, according to site's standard practice) with or without hormonal therapy (mandatory if positive hormone receptors). Participants will be followed for up to 5 years from start of neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants with early stage HER2-positive breast cancer
* Scheduled to receive neoadjuvant therapy with the objective of conservative surgery
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2

Exclusion Criteria:

* Participants with partial or total lobular carcinoma
* Participants with inflammatory breast cancer
* Previous treatment with chemotherapy, radiation therapy or hormonal therapy for breast cancer
* Previous history of cancer (other than curatively treated basal and squamous cell carcinoma of the skin and/or in situ carcinoma of the cervix) relapsing within the 5 years before study entry or in situ contralateral breast carcinoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2010-05-19 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Pathological Complete Response as per Chevallier's Classification as Reviewed by an Independent Committee | After 6 cycles (18 weeks) of neoadjuvant therapy (cycle length=21 days)

SECONDARY OUTCOMES:
Percentage of Participants With Pathological Complete Response According to Chevallier's Classification as per Local Procedures | After 6 cycles (18 weeks) of neoadjuvant therapy (cycle length=21 days)
Percentage of Participants With Pathological Complete Response According to Sataloff's Classification as Reviewed by an Independent Committee | After 6 cycles (18 weeks) of neoadjuvant therapy (cycle length=21 days)
Percentage of Participants With Ultrasound Response According to Modified Response Evaluation Criteria in Solid Tumors (RECIST) | Neodajuvant treatment period (21 weeks)
Percentage of Participants With Conservative Surgery Post Neoadjuvant Treatment | Week 20 (between Day 28 and Day 35 after the Cycle 6, cycle length=21 days)
Local Relapse-Free Interval (LRFI) According to Modified RECIST Criteria | From baseline to occurrence of relapse/disease or death of any cause (up to 5 years)
Disease-Free Survival (DFS) According to Modified RECIST Criteria | From baseline to occurrence of relapse/disease or death of any cause (up to 5 years)
Distant Disease-Free Interval (DDFI) According to Modified RECIST Criteria | From baseline to occurrence of relapse/disease or death of any cause (up to 5 years)
Overall Survival | Baseline up to occurrence of death (up to 5 years)
Percentage of Participants With Adverse Events | Baseline up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (28):
- France (28):
  - Centre Radiotherapie Marie Curie, Arras
  - Centre Hospitalier; Hematologie-Oncologie, Beauvais
  - Clinique Tivoli; Sce Radiotherapie, Bordeaux
  - Hopital Augustin Morvan; Federation De Cancerologie, Brest
  - Centre Jean Perrin; Hopital De Jour, Clermont-Ferrand
  - Pole Sante Republique;Oncologie Hematologie, Clermont-Ferrand
  - Centre Georges Francois Leclerc; Oncologie 3, Dijon
  - Institut Daniel Hollard, Grenoble
  - Centre Hospitalier Departemental Les Oudairies, La Roche-sur-Yon
  - Hopital Dupuytren; Oncologie Medicale, Limoges
  - Centre Leon Berard; Oncologie Genetique, Lyon
  - Hopital Clinique Claude Bernard; Oncologie Medicale, Metz
  - Ch De Montlucon; Sce Med Interne Hemato Onco, Montluçon
  - Institut régional du Cancer Montpellier, Montpellier
  - Centre D'Oncologie de Gentilly; Oncology, Nancy
  - Centre Antoine Lacassagne; Hopital De Jour A2, Nice
  - Institut Curie; Oncologie Medicale, Paris
  - GH Paris Saint Joseph; Hopital De Jour Oncologie, Paris
  - HOPITAL TENON; Cancerologie Medicale, Paris
  - Clinique Francheville; Radiotherapie, Périgueux
  - Institut Jean Godinot; Oncologie Medicale, Reims
  - Centre Eugene Marquis; Unite Huguenin, Rennes
  - Clinique de L'Union; Oncologie, Saint-Jean
  - Institut de Cancerologie de La Loire; Radiotherapie, Saint-Priest-en-Jarez
  - Centre Paul Strauss; Oncologie Medicale, Strasbourg
  - Clinique Pasteur; Oncologie Medicale, Toulouse
  - Centre Henry S Kaplan - CHU Bretonneau ; service oncologie, Tours
  - Centre Alexis Vautrin; Oncologie Medicale, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Coudert B, Pierga JY, Mouret-Reynier MA, Kerrou K, Ferrero JM, Petit T, Kerbrat P, Dupre PF, Bachelot T, Gabelle P, Giard S, Coeffic D, Bougnoux P, Prevost JB, Paintaud G, Thibault G, Hernandez J, Coudert M, Arnould L, Berriolo-Riedinger A. Use of [(18)F]-FDG PET to predict response to neoadjuvant trastuzumab and docetaxel in patients with HER2-positive breast cancer, and addition of bevacizumab to neoadjuvant trastuzumab and docetaxel in [(18)F]-FDG PET-predicted non-responders (AVATAXHER): an open-label, randomised phase 2 trial. Lancet Oncol. 2014 Dec;15(13):1493-1502. doi: 10.1016/S1470-2045(14)70475-9. Epub 2014 Oct 30. PMID 25456368